CLINICAL TRIAL: NCT05144555
Title: Periodontal Evaluation in Patients Undergoing Fixed Orthodontic Treatment With Stainless Steel or Ceramic Brackets: a Clinical Trial.
Brief Title: Periodontal Parameters in Orthodontic Patients With Stainless Steel and Ceramic Brackets.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Research Resident, Principal Investigator, University of Pavia
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2021-METCERIGIENE
Record Dates: First submitted 2021-11-20; First posted 2021-12-03 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Periodontal Inflammation; Dental Malocclusion
Keywords: orthodontic brackets; ceramic brackets; stainless steel brackets; orthodontic fixed treatment; dental hygiene
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group MET (Experimental): Patients from this group will undergo orthodontic fixed treatment with stainless steel brackets.
  Interventions: Other: Fixed orthodontic treatment with stainless steel brackets
- Group CER (Active Comparator): Patients from this group will undergo orthodontic fixed treatment with ceramic brackets.
  Interventions: Other: Fixed orthodontic treatment with ceramic brackets

INTERVENTIONS:
Other: Fixed orthodontic treatment with stainless steel brackets — Stainless steel brackets (Queen Series Low Profile Brackets MBT 0.022", Aestetika, Terni, TR, Italy) will be applied on the vestibular surfaces of teeth to perform orthodontic treatment.
  Arms: Group MET
Other: Fixed orthodontic treatment with ceramic brackets — Ceramic brackets (Super Clear Series Brackets MBT 0.022", Aestetika, Terni, TR, Italy) will be applied on the vestibular surfaces of teeth to perform orthodontic treatment.
  Arms: Group CER

SUMMARY:
The aim of this study is to assess if there are significant differences in periodontal conditions between patients undergoing fixed orthodontic treatment with stainless steel or ceramic brackets. For this study, patients will be enrolled and divided into two groups, according to the type of brackets (stainless steel or ceramic) used for orthodontic treatment. A professional supragingival and subgingival oral hygiene will be performed before the bonding of the orthodontic brackets together with a periodontal evaluation will be recording the following periodontal indices: PPD, BoP, BS, GI, PI, BEWE and Schiff Air Index. Indices will be recorded after 1, 3 and 6 months after the bonding, separately for both in maxillary and in mandibular dental arches and only for teeth with brackets bonded.

DETAILED DESCRIPTION:
This clinical trial aims to investigate if there are significant differences in periodontal conditions between patients undergoing fixed orthodontic treatment with stainless steel or ceramic brackets. Patients recruited for the study will be asked to sign the informed consent. Parents will sign the consent for underage patients. A professional supragingival and subgingival oral hygiene will be performed before the bonding of the orthodontic brackets; a piezoelectric instrument and Gracey curettes will be used. After that, patients will be divided into two groups:

* Group MET: stainless steel brackets will be bonded on the vestibular surfaces of teeth.
* Group CER: ceramic brackets will be bonded on the vestibular surfaces of teeth. Before the bonding on maxillary dental arch, a periodontal evaluation will be conducted recording the following periodontal indices: PPD, BoP, BS, GI, PI, BEWE and Schiff Air Index. Indices will be recorded after 1, 3 and 6 months after the bonding, separately for both in maxillary and in mandibular dental arches. Only teeth with brackets bonded will be considered.

ELIGIBILITY:
Inclusion Criteria:

* patients willing to begin fixed multibracket therapy with metallic or ceramic brackets;
* full permanent dentition;
* all teeth from central incisors to second premolars.

Exclusion Criteria:

* patients suffering from systemic diseases;
* patients taking medications that could alter periodontal conditions (NSAIDS, steroids, etc.);
* patients with low compliance;
* patients unable to give informed consent;
* presence of congenital enamel defects;
* extractions for orthodontic reasons;
* oral/orthognathic surgery;
* presence of dental implants on teeth from central incisors to second premolars.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-12-18 (Actual); Primary Completion 2024-09-09 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
Change in GI - Gingival Index (Loe and Silness, 1963) | Before the bonding procedure; after 1, 3 and 6 months after the bonding both in maxillary and in mandibular dental arches
  Scoring criteria:
  * 0 = normal gingiva
  * 1 = mild inflammation, edema and swelling; no bleeding
  * 2 = moderate inflammation with edema, swelling and bleeding on probing
  * 3= severe inflammation with marked edema, redness, tissues, ulceration and spontaneous bleeding
Change in BS - Bleeding Score | Before the bonding procedure; after 1, 3 and 6 months after the bonding both in maxillary and in mandibular dental arches
  Scoring criteria:
  * 0 = no bleeding
  * 1 = punctiform bleeding in the site of probing
  * 2 = slightly extended bleeding in the site of probing
  * 3 = bleeding in more than a half of gingival margin
  * 4= gingival border fully covered by blood
Change in PI - Plaque Index (Silness and Löe, 1964) | Before the bonding procedure; after 1, 3 and 6 months after the bonding both in maxillary and in mandibular dental archesBefore the bonding procedure; after 1, 3 and 6 months after the bonding both in maxillary and in mandibular dental arches
  Scoring criteria:
  * 0 = no plaque
  * 1 = thin plaque layer at the gingival margin, only detectable by scraping with a probe
  * 2 = moderate layer of plaque along the gingival margin; interdental spaces free, but plaque is visible to the naked eye
  * 3= abundant plaque along the gingival margin; interdental spaces filled with plaque
Change in BEWE index (Basic Erosive Wear Examination) | Before the bonding procedure; after 1, 3 and 6 months after the bonding both in maxillary and in mandibular dental archesBefore the bonding procedure; after 1, 3 and 6 months after the bonding both in maxillary and in mandibular dental arches
  Scoring criteria:
  * 0 = no ETW (erosive tooth wear)
  * 1 = initial loss of surface texture
  * 2 = distinct defect; hard tissue loss involving <50% of the surface area
  * 3 = hard tissue loss involving ≥50% of the surface area
Change in Schiff Air Index - sensitivity score | Before the bonding procedure; after 1, 3 and 6 months after the bonding both in maxillary and in mandibular dental archesBefore the bonding procedure; after 1, 3 and 6 months after the bonding both in maxillary and in mandibular dental arches
  Evaluation criteria with the visual analog scale (VAS). The patient indicates the pain level on the scale of 0-10
Change in PPD - Probing Pocket Depth | Before the bonding procedure; after 1, 3 and 6 months after the bonding both in maxillary and in mandibular dental archesBefore the bonding procedure; after 1, 3 and 6 months after the bonding both in maxillary and in mandibular dental arches
  Evaluation (in mm) of the depth of the gingival sulcus, through a millimeter periodontal probe; it is detected from the gingival margin to the bottom of the gingival sulcus or periodontal pocket, evaluated at 6 sites.
Change in BOP - Bleeding on Probing (percentage) | Before the bonding procedure; after 1, 3 and 6 months after the bonding both in maxillary and in mandibular dental archesBefore the bonding procedure; after 1, 3 and 6 months after the bonding both in maxillary and in mandibular dental arches
  Site-specific assessment of the presence or absence of gum bleeding after the insertion of the periodontal probe. Percentage of sites with bleeding on probing determines the BOP%.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, DDS, PhD, Principal Investigator — University of Pavia
Locations (1):
- Unit of Orthodontics and Pediatric Dentistry - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Pediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available upon motivated request to Principal Investigator.